CLINICAL TRIAL: NCT06520228
Title: Effects of Active Video Games on Motor Coordination of Early Childhood--Focusing on Children in Zhengzhou, China
Brief Title: The Purpose of This Study is to Reveal the Influence of Active Video Games on Children's Motor Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Lu Chenxi, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024109
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: The Study Demonstrated the Effect of Active Video Games on Motor Coordination in Children Over a 12-week Intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active video games (Experimental)
  Interventions: Behavioral: Active video games
- Traditional sports games (Experimental)
  Interventions: Behavioral: Traditional sports games

INTERVENTIONS:
Behavioral: Active video games — The experiment was divided into two groups. One experimental group, one control group. The experimental group received an active video game intervention for 12 weeks, 40 minutes twice a week. The control group underwent 12 weeks of traditional physical activity, 40 minutes twice a week.
  Arms: Active video games
Behavioral: Traditional sports games — The experiment was divided into two groups. One experimental group, one control group. The experimental group received an active video game intervention for 12 weeks, 40 minutes twice a week. The control group underwent 12 weeks of traditional physical activity, 40 minutes twice a week.
  Arms: Traditional sports games

SUMMARY:
The goal of the study was to understand the effects of active video games on motor coordination in children. The main questions it aims to answer are:

The effect of positive video games on children's motor ability.

Researchers will compare traditional physical activities to see if active video games are effective in improving motor coordination in children.

Participants will:

Play active video games twice a week for 12 weeks Data were collected during the first and twelfth weeks

ELIGIBILITY:
Inclusion Criteria:

1. Children who meet the age requirements；
2. Have basic language skills;
3. Not require medication;
4. The parents agrees to participate.

Exclusion Criteria:

1. Those with the eye, ear, or physical disabilities or other physical health problems that prevent them from participating in training.
2. Those with severe organic diseases of the heart, liver, kidneys, and other organs
3. Patients with severe central system pathology.
4. Patients with acute infectious diseases, Etc., who are not suitable to participate in training.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
baseline | The first week of the experiment.
  The subjects (control group and experimental group) will be pre-tested during the first week of the experiment. The motor coordination ability of the subject was obtained. Motor coordination was measured using the Motor Assessment Battery for Children - Second Edition (MABC-2).

SECONDARY OUTCOMES:
post test1 | The 12th week of the experiment.
  The subjects (control group and experimental group) will be tested after the 12th week of the experiment. The motor coordination ability of the subject was obtained. Motor coordination was measured using the Motor Assessment Battery for Children - Second Edition (MABC-2).

CONTACTS AND LOCATIONS:
Locations (1):
- Lu Chenxi, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No